CLINICAL TRIAL: NCT06526286
Title: Clinical Decision Support to Increase Use of Medications for Opioid Use Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-1188; 24-1188 (Other: IRB protocol); R61DA057610 (NIH)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Medication Abuse; Harm Reduction; Opioid Use Disorder; Supportive Care
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction; Opioid-Related Disorders | interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Control group to enable tracking of temporal changes in prescribing. Providers will not see any alert.
- CDS Notification: Providers will see a clinical decision support tool within the electronic health record when treating a patient at risk for opioid use disorder to encourage the provider to use a clinical care pathway to assess for opioid use disorder and when applicable, treat opioid use disorder with buprenorphine. Smart text will also be available in the electronic health record so that the provider can easily document screening and treatment discussions with the patient.
  Interventions: Other: Medications for Opioid Use Disorder Pathway Clinical Decision Support (CDS)

INTERVENTIONS:
Other: Medications for Opioid Use Disorder Pathway Clinical Decision Support (CDS) — Clinical decision support (CDS) in the form of an electronic health record (EHR)-integrated, provider-facing notification suggesting (a) the patient may be at risk for opioid use disorder and could benefit from screening, (b) patients with opioid use disorder would benefit from treatment with buprenorphine and (c) utilization of a clinical care pathway to help treat patients with opioid use disorder with buprenorphine as suggested by the Center for Disease Control and Prevention (CDC) guidelines.
  Groups: CDS Notification

SUMMARY:
The objective of this study is to evaluate the impact of clinical decision support (CDS) in the form of an alert to identify patients who may be at risk of opioid use disorder (OUD) and a clinical care pathway helping providers treating patients with opioid use disorder. The pathway provides health care providers with information and suggestions for screening and treatment of opioid use disorder, including treatment with medications. The 2022 Centers for Disease Control and Prevention (CDC) clinical practice guideline for prescribing opioids for pain recommends providers asses for and treat opioid use disorder using approved medications for opioid use disorder (MOUD). This project will randomize primary care providers at the clinic level to a control arm or intervention arm. The control arm will have access to the clinical care pathway, but will not be reminded to utilize the pathway when treating a patient with opioid use disorder. The intervention arm will receive a reminder nudge about the pathway. Buprenorphine (a medication used to treat opioid use disorder) prescribing behavior of providers and outcomes of patients will be examined based on medical records data collected during routine care. The study period will be approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary care encounter AND
* Current opioid prescription (not buprenorphine) and Active opioid medications over the last 90 days OR
* Documented as on local Pain Registry "Does the patient fit the criteria to be included on the Pain Registry?" OR
* Has active problem list diagnosis of long-term (current) use of opiate analgesic OR
* Is taking >=90 morphine milligram equivalents (MME) per day OR
* Prior positive toxicology screen for illicit drugs OR
* Diagnosis of opioid use disorder

Exclusion Criteria:

* Active cancer diagnosis in the last 1 year
* Hospice care/palliative care order
* Sickle cell disease diagnosis

Ages: 12 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents and visitors to the state of Colorado who seek healthcare within the University of Colorado Health (UCHealth) primary care system.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients at risk for opioid use disorder receiving medications for opioid use disorder | 18 months
  The number of primary care patients identified to be at risk for opioid use disorder treatment with buprenorphine for treatment divided by the total number of patients meeting opioid use disorder criteria

SECONDARY OUTCOMES:
Clinical decision support (CDS) acceptance rate | 18 months
  The number of times providers accepted the clinical decision support (CDS) tool and utilized the clinical care pathway in treating opioid use disorder.
Subsequent opioid overdose/poisoning rates | Six months after an encounter where the opioid use disorder is identified
  The number of patients who had a diagnosis of opioid overdose or poisoning
Buprenorphine initiation | Six months after an encounter where the opioid use disorder is identified
  Number of patients who filled a buprenorphine prescription after being identified at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hoppe, DO, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: Yes
De-identified data utilized in this project will be housed on the National Addiction and HIV Data Archive Program (NAHDAP) after results of the study are published.
Supporting Information: Study Protocol
Time Frame: Data will be provided to National Addiction and HIV Data Archive Program (NAHDAP) after study results are published in peer-reviewed journals.
Access Criteria: Prior to downloading study data, the individual will have to register with the site and agree to a standard data use agreement
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/